CLINICAL TRIAL: NCT01620541
Title: Comparing Ankle Arthrodesis to Ankle Arthroplasty
Brief Title: Comparing Ankle Fusion to Ankle Replacement
Status: Active, not recruiting | Type: Observational
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Institutes of Health (NIH) (NIH); University of Washington (Other); Orthopedic + Fracture Specialists, Portland, OR (Other); Minnesota Orthopedic Sports Medicine Institute at Twin Cities Orthopedics (Unknown); Orthopaedic and Spine Center of the Rockies (Unknown); Orthopaedic Associates of Michigan, PC (Other)
Responsible Party: Sponsor
Other Study IDs: SB223; 1R01AR056316-01A2 (NIH)
Record Dates: First submitted 2012-06-11; First posted 2012-06-15 (Estimated); Last update posted 2025-04-08 (Actual); Status verified 2024-04

CONDITIONS: End-stage Ankle Arthritis (ESAA); Osteoarthritis (OA)
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Ankle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Preference, Ankle Arthrodesis
  Interventions: Procedure: Ankle Arthrodesis
- Preference, Ankle Arthroplasty
  Interventions: Procedure: Ankle Arthroplasty

INTERVENTIONS:
Procedure: Ankle Arthrodesis — All surgeons will employ a well-established technique of rigid internal fixation. In this technique, the joint is prepared by removing cartilage from the surfaces, the bones are positioned as desired, and screws and/or a plate are attached to compress the bones together and prevent motion. This technique obviates the need for a cast or external support. Patients are allowed to walk with weight bearing aids immediately. Radiographs are performed at 6 weeks to determine weight bearing status. Weight is allowed on the limb in increments over the 6 to 12 weeks after surgery.
  Other Names: Ankle Fusion
  Groups: Preference, Ankle Arthrodesis
Procedure: Ankle Arthroplasty — Protocols are similar among participating centers. Each surgeon uses an anterior surgical approach between the tibialis anterior tendon and the toe extensor group, splints the ankles for 2 weeks, and restricts weight bearing for the first 6 weeks. Radiographs are performed at 6 weeks to determine weight bearing status. The study involves only FDA approved implants with which the surgeon has established experience.
  Other Names: Total Ankle Replacement
  Groups: Preference, Ankle Arthroplasty

SUMMARY:
End-stage ankle arthritis (ESAA) is a debilitating condition associated with severe pain, dysfunction, and reduced quality of life. Many patients with ESAA have difficulty walking for even 100 feet or up a single flight of stairs. Patients seeking surgery for ESAA have two primary treatment options: ankle arthrodesis (i.e., ankle fusion) and ankle arthroplasty (i.e., ankle replacement). Few studies have directly compared the effectiveness of these two procedures, and no randomized controlled trials (RCTs) have been performed.

The investigators will compare the following in subjects undergoing ankle arthrodesis and ankle arthroplasty before surgery, and post-surgery at 3 and 6 months, and on an annual basis up to ten years.

1. Overall physical function and ankle specific function
2. Ankle pain intensity and interference with activities
3. Activity levels
4. Overall general health
5. Post-surgical complication rates

The investigators will also identify prognostic factors that are predictive of higher physical function, ankle specific function, reduced pain, improved general health, and overall patient satisfaction.

DETAILED DESCRIPTION:
From study inception until March 2014, the investigators conducted a multi-site randomized controlled trial (RCT) comparing the effectiveness of ankle arthrodesis and ankle arthroplasty over a 2-year follow-up period. The study used a modified Comprehensive Cohort Design. Subjects unwilling to randomize to surgery could still participate in the study by entering into the preference cohort and select surgery in consultation with their surgeon.

By March 2014, no subjects had entered into the randomized cohort. The Data and Safety Monitoring Board (DSMB) recommended stopping recruitment in the randomized arm of the study since no subjects were willing to randomize to surgery. All patients were enrolled in the preference cohort and selected arthrodesis or arthroplasty. Despite the change in study design, the objectives remain unchanged.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ankle arthritis
2. Failed conservative care and deemed a surgical candidate
3. Adult patients between 21 and 89 years of age
4. Ambulatory but whose primary impediment to pain-free ambulation is ankle arthritis

Exclusion Criteria:

1. Recent surgical, neurological, metabolic, or lower limb musculoskeletal problem that might impair the ambulation measures in the study such as severe knee or hip osteoarthritis
2. Complicated procedures requiring multiple corrections
3. Inflammatory arthritis with multi-focal disease (i.e. arthritis that affects multiple parts of the body)
4. Inadequate cognitive or language function to consent to participate
5. Unable or unwilling to participate in clinic follow-ups and/or remote follow-ups for 24 months after surgery
6. Unwilling or unable to comply with postoperative management program
7. Lack of a telephone number or stable mailing address

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are recruited from surgical foot and ankle orthopedic clinics at the participating study sites.
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in overall physical function and ankle specific function between subjects undergoing ankle arthrodesis and total ankle arthroplasty | Before surgery, and post-surgery at 3 and 6 months, and on an annual basis up to ten years.
  Questionnaire data (Foot and Ankle Ability Measure; SF-36 Health Survey)
Change in overall pain intensity and ankle specific pain intensity; Interference with activities in subjects undergoing ankle arthrodesis and total ankle arthroplasty | Before surgery and post-surgery at 3 and 6 months, and on an annual basis up to ten years.
  Questionnaire data (Foot and Ankle Ability Measure; Chronic Pain Grade)
Change in general health in subjects undergoing ankle arthrodesis and total ankle arthroplasty | Before surgery and post-surgery at 3 and 6 months, and on an annual basis up to ten years.
  Questionnaire data (Functional Comorbidity Index and SF-36 Health Survey)

SECONDARY OUTCOMES:
Intrinsic and extrinsic prognostic factors which are predictive of higher physical function, ankle specific function, reduced pain, improved general health, and overall patient satisfaction | Assessed before surgery and post-surgery at 3 and 6 months, and on an annual basis up to ten years.
  Medical record review and questionnaire data
Post-surgical complication rates | Assessed monthly until 24 months after surgery
  Medical record review
Change in daily step counts | Before surgery and at 6, 12, and 24 months after surgery
  Step counts using a StepWatch Activity Monitor, worn for a 7-14 day time period.
Change in patient satisfaction | Done post-surgery at 3 and 6 months, and on an annual basis up to ten years.
  Questionnaire data

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J Sangeorzan, MD, Principal Investigator — VA Puget Sound Health Care System & University of Washington
Locations (6):
- United States (6):
  - Orthopaedic and Spine Center of the Rockies, Fort Collins, Colorado
  - Orthopaedic Associates of Michigan, Grand Rapids, Michigan
  - Twin Cities Orthopedics, Edina, Minnesota
  - Orthopedic + Fracture Specialists, Portland, Oregon
  - Harborview Medical Center, Seattle, Washington
  - VA Puget Sound Health Care System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No